CLINICAL TRIAL: NCT03007680
Title: Effect of Core Muscles Activation for the Increase of Quality in Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Wonhee Kim, Assistant Professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HURF-2016-44
Record Dates: First submitted 2016-12-30; First posted 2017-01-02 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Core muscle activation (Experimental): Core muscle will be activated by physical fitness using plank, crunch and leg extension.
  Interventions: Other: Core muscle activation
- No core muscle activation (No Intervention)

INTERVENTIONS:
Other: Core muscle activation
  Arms: Core muscle activation

SUMMARY:
The purpose of this study is to determine whether core muscle activation is effective in the increase of quality of cardiopulmonary resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses who have experiences of CPR education

Exclusion Criteria:

* 1. Acute/chronic pain on body 2. History of cardiovascular disease 3. History of vertebral disease including herniated disc 4. Pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
chest compression depth | 4 min
lean depth | 4 min
high quality chest compressions | 4 min
  frequency of chest compressions satisfying the condition that 5-6cm chest compression depth and lean depth less than 2mm
chest compressions rate | 4 min

SECONDARY OUTCOMES:
elbow angle | 4 min
  measured by motion sensor during chest compressions
muscle fatigue | 4 min
  measured by EMG during chest compressions

CONTACTS AND LOCATIONS:
Overall Officials: Wonhee Kim, M.D., Principal Investigator — Hallym University
Locations (1):
- Hallym University Kangnam Sacred Hospital, Seoul, South Korea